CLINICAL TRIAL: NCT02839681
Title: Phase II Trial With Safety Run-in of the Anti-Mesothelin Antibody Drug Conjugate Anetumab Ravtansine for Mesothelin Expressing Lung Adenocarcinoma
Brief Title: Anti-Mesothelin Antibody Drug Conjugate Anetumab Ravtansine for Mesothelin Expressing Lung Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow, insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160145; 16-C-0145
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Lung Neoplasms
Keywords: Lung Adenocarcinoma; Immunotoxin; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung | interventions — anetumab ravtansine; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- 1/Safety Run-in Arm (Experimental): Subjects will be dosed with the higher of the 2 possible anetumab ravtansine doses (dose level 1) evaluated on the study
  Interventions: Drug: Anetumab Ravtansine; Device: Blood test
- 2/Phase 2 Arm (Experimental): Subjects will be dosed with anetumab ravtansine at the recommended phase 2 dose (dose level 1 if no more than 1 dose limiting toxicity (DLT) occurred in the safety run-in arm, or at dose level -1 otherwise)
  Interventions: Drug: Anetumab Ravtansine; Device: Blood test

INTERVENTIONS:
Drug: Anetumab Ravtansine — Administered intravenously (IV) every 3 weeks
  Other Names: BAY 94-9343
Device: Blood test — Research blood test for eligibility

SUMMARY:
Background:

Anetumab ravtansine is a new drug. It kills cancer cells that carry mesothelin. That is a protein on the surface of tumor cells in many types of tumors, including most lung cancers. Researchers want to find a safe dose for the study drug for lung cancer. They want to see if it can shrink tumors in mesothelin-positive lung cancer.

Objectives:

To test the safety and effectiveness of anetumab ravtansine for lung cancer.

Eligibility:

Adults 18 years and older who have lung cancer that has gotten worse on other therapy

Design:

Participants will be screened with:

Medical history

Physical exam

Tumor tissue sample. This can be from a previous procedure.

Blood and urine tests

Heart tests

Scans. For one scan, a small amount of radioactive substance is injected into the blood.

Eye exam

The study will have 21-day cycles.

On day 1 of each cycle, participants will get the study drug through a tube inserted in a vein.

Participants will repeat a heart test in cycles 1 and 2.

They will have blood tests weekly in cycle 1, twice in all other cycles.

They will have scans every 6 weeks for the first 6 months, every 9 weeks until the end of year 2, then every 12 weeks.

Participants will have samples of tumor tissue taken twice.

About 30 days after stopping the study drug, participants will have a follow-up visit. This will include medical history, physical exam, blood and pregnancy tests, and heart and eye tests.

Some will be called a few times a year to discuss their health and treatment.

DETAILED DESCRIPTION:
Background:

* Lung cancer is the leading cause of cancer-related death worldwide, accounting for more than one million deaths every year.
* Non-small-cell lung cancer (NSCLC) constitutes approximately 85% of lung cancers and about 40% of patients with newly diagnosed NSCLC have advanced disease. The median year overall survival for advanced NSCLC is at least 1 year.
* In recent years, identification of oncogenic alterations such as mutations in epidermal growth factor receptor (EGFR) and anaplastic large-cell lymphoma kinase (ALK) translocations and therapies targeting tumor immune escape mechanisms have led to a substantial improvement in the prognosis of patients with advanced lung cancer;

however, such alterations have been detected in less than half of all advanced NSCLC patients in only a small subset of patients respond to immunotherapeutic interventions available today.

* Anetumab ravtansine (BAY 94-9343) is an antibody-drug conjugate targeting mesothelin, a protein normally present on mesothelial cells. A Phase I trial showed the overall acceptable and manageable safety profile. It is being developed for patients with mesothelin expressing cancers; clinical development is furthest along in mesothelioma where it is in a registration phase II clinical trial.
* National Cancer Institute (NCI) researchers have demonstrated that mesothelin messenger ribonucleic acid (mRNA) and protein are present in a substantial number of lung adenocarcinoma cell lines; mesothelin expression has been observed in over 50% of advanced lung adenocarcinomas by immunohistochemical assessment.

Objectives:

Safety Run-in

-To evaluate safety and tolerability of anetumab ravtansine in patients with previously treated unresectable mesothelin expressing advanced lung adenocarcinoma (stage IIIB or IV).

Phase 2

-To determine the efficacy (objective response rate) of anetumab ravtansine in patients with advanced (Stage IIIb) or metastatic (Stage IV) mesothelin expressing lung adenocarcinoma.

Eligibility:

* Age >18 years.
* Histologically or cytologically confirmed previously treated unresectable mesothelin expressing advanced lung adenocarcinoma (stage IIIB or IV)
* Positive mesothelin expression in the archival tumor tissue, defined as the mesothelin membrane intensity score of 2+ or 3+ (on the 0-3 scale) expressed on the membrane of greater than or equal to 10% of tumor cells.
* Should have received at least one prior platinum based chemotherapy and an immune checkpoint targeted agent. In addition, subjects with epidermal growth factor receptor [EGFR]-mutated and anaplastic lymphoma kinase [ALK]-translocated NSCLC should have received Food and Drug Administration (FDA)-approved targeted therapies as appropriate.
* Normal organ function

Design:

* This is an open label, single center, phase I/II study of anetumab ravtansine in subjects with mesothelin positive lung adenocarcinoma.
* During the safety run-in portion of the study, de-escalating doses will be assessed to determine a recommended phase 2 dose (RP2D).
* During the phase 2 portion of the study, the (RP2D) will be assessed for objective response rate.
* During both portions of the study, anetumab ravtansine will be administered intravenously every 3 weeks until disease progression in the absence of clinical benefit, patient withdrawal or the occurrence of intolerable toxicities.
* Response assessments (imaging) will occur every 6 weeks for the first 6 months, then every 9 weeks until the end of year 2, then every 12 weeks thereafter.
* Up to 12 evaluable patients will be enrolled in the safety run-in portion of the study. Approximately twenty patients, including 6 from the safety run-in portion of the study, will be evaluated in the phase 2 portion of the study. The accrual ceiling will be set at 55 to accommodate screen failures (a 50% failure rate with regard to mesothelin expression) and inevaluable subjects.

ELIGIBILITY:
* INCLUISION CRITERIA:

Subjects must have histologically or cytologically confirmed previously treated unresectable mesothelin expressing advanced lung adenocarcinoma (stage IIIB or IV) as confirmed by the Laboratory of Pathology, National Cancer Institute (NCI)

Subjects must have positive mesothelin expression in the archival tumor tissue, defined as the mesothelin membrane intensity score of 2+ or 3+ (on the 0-3 scale) expressed on the membrane of greater than or equal to 10% of tumor cells.

Subjects must provide sample of archival tumor tissue (tissue block preferred, at least 5 formalin-fixated, paraffin-embedded [FFPE] slides acceptable) collected any time before the general screening. A fresh biopsy will be collected if archival sample is unavailable or insufficient.

Subjects must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan. See Section 6.3 for the evaluation of measurable disease.

Subjects with resected primary tumors who have documented metastases are eligible.

Subjects should have received at least one prior platinum based chemotherapy and an immune checkpoint targeted agent. Subjects with epidermal growth factor receptor [EGFR]-mutated and anaplastic lymphoma kinase [ALK]-translocated non-small cell lung cancer (NSCLC) should have received Food and Drug Administration (FDA)-approved targeted therapies as appropriate.

Age >18 years. Because no dosing or adverse event data are currently available on the use of anetumab ravtansine in subjects <18 years of age, children are excluded from this study.

Eastern Cooperative Oncology Group (ECOG) performance status < or equal to 2

Subjects must have adequate bone marrow function as assessed by the following laboratory test results:

* Hemoglobin greater than or equal to 9.0 g/dL or greater than or equal to 5.6 mmol/L
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3 or greater than or equal to 1.5 x 10^9/L
* Platelet count greater than or equal to 100,000/mm^3 or greater than or equal to 100 x 10^9/L

Subjects must have adequate kidney function, with serum creatinine <1.5 x ULN or calculated glomerular filtration rate (GFR) of > 45/mL/min/1.73 m^2

Subjects must have adequate liver function as assessed by the following laboratory test results:

* Total bilirubin less than or equal to 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 3.0 times upper limit of normal (ULN) in subjects without liver metastases or 5.0 times ULN in subjects with liver metastases

Subjects must have adequate coagulation, as assessed by the following laboratory test results:

* International normalized ratio (INR) or prothrombin time (PT) less than or equal to 1.5 x ULN
* Partial thromboplastin time (PTT) less than or equal to 1.5 x ULN

Due to the lack of adequate reproductive toxicity data on anetumab ravtansine, subjects must use 2 forms of highly effective contraception concomitantly from the initiation of study therapy until 6 months after the last dose of study therapy. Additionally, the use of condoms is required. It should also be noted that, where 2 forms of effective contraception are required, a subject may choose to use a double-barrier method consisting of condom and cervical occlusive cap / diaphragm with spermicide

Ability of subject to understand and the willingness to sign a written informed consent document.

Subjects must provide a signed informed consent before any screening procedures.

EXCLUSION CRITERIA:

Subjects who have a previous or concurrent cancer that is distinct in primary site or histology from lung adenocarcinoma, except cervical carcinoma in situ, treated basal cell carcinoma, superficial noninvasive bladder tumors or any previous cancer curatively treated <2 years before the start of study treatment.

Subjects who have a history or current evidence of bleeding disorder, i.e. any hemorrhage/bleeding event of Common Terminology Criteria in Adverse Events (CTCAE) Grade greater than or equal to 2 within 4 weeks before the start of study treatment.

History of symptomatic metastatic brain or meningeal tumors unless the subject is > 3 months from definitive therapy and has no evidence of tumor growth on an imaging study within 2 weeks prior to study entry. Subjects with brain metastases must not be undergoing acute corticosteroid therapy or steroid taper. Chronic steroid therapy is acceptable provided that the dose is stable for one month prior to screening.

Subjects who have a history or current evidence of uncontrolled cardiovascular disease including but not limited to the following conditions:

* Congestive heart failure of New York Heart Association (NYHA) Class III or IV
* Unstable angina (symptoms of angina at rest) or new-onset angina within <3 months before the start of study treatment.
* Arterial thrombosis, deep vein thrombosis, or pulmonary embolism within <3 months before the start of study treatment.
* Myocardial infarction or stroke within <3 months before the start of study treatment.
* Pericarditis (any CTCAE grade), pericardial effusion (CTCAE Grade greater than or equal to 2) or pleural effusion (CTCAE Grade greater than or equal to 2)
* Cardiac arrhythmia requiring anti-arrhythmic therapy. Subjects receiving digoxin, calcium channel blockers except verapamil, or beta-adrenergic blockers except propranolol are eligible at the investigators discretion if the dose has been stable for at least 2 weeks before the start of study treatment. Subjects with sinus arrhythmia and infrequent premature ventricular contractions are eligible at the investigators discretion.

Subjects who have a left ventricular ejection fraction (LVEF) <50%, as assessed by echocardiogram performed at screening.

Subjects who have a corrected Q wave, T wave (QT) (corrected QT interval by Fredericia (QTcF)) interval >480 ms (CTCAE Grade >1) determined by the electrocardiogram (ECG) recorders algorithm on the screening ECG.

Subjects who have a history or current evidence of uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg at screening despite optimal medical management. Subjects with a history of mild to moderate

hypertension are eligible at the investigator s discretion if the hypertension is adequately controlled by antihypertensive treatment used at a stable dose for at least 2 weeks before the start of study treatment.

Subjects who have a heart rate greater than or equal to 100 beats per minute (bpm) or less than or equal to 45 bpm determined by the ECG recorder s algorithm on the screening ECG.

Women who are pregnant or breast-feeding. Women of reproductive potential must have a negative serum beta human chorionic gonadotropin (beta-HCG) pregnancy test obtained within 7 days before the start of study treatment.

Subjects who have had a major surgery or significant trauma within 4 weeks before the start of study treatment.

Subjects who have had solid organ or bone marrow transplantation.

Subjects who have a history of hypersensitivity to any of the study drugs or their excipients, or a history of severe hypersensitivity to any other antigen.

Subjects who have a history of human immunodeficiency virus (HIV) infection or subjects who have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection. Subjects with chronic HBV or HCV infection are eligible at the investigators discretion if the subject is considered non-infectious based on serological markers.

Subjects who have an active clinically serious infection of CTCAE Grade greater than or equal to 2.

Subjects with a non-healing serious wound, ulcer, or bone fracture unrelated to the primary tumor.

Subjects with corneal epitheliopathy or any eye disorder that may predispose the subjects to drug-induced corneal epitheliopathy, or may interfere with diagnosis of treatment-emergent corneal epitheliopathy at the discretion of the investigator in consultation with the ophthalmologist/optometrist. Low grades of superficial punctate keratitis, within the range seen in the normal population, should not lead to the exclusion of the patient

Subjects experiencing unresolved toxicity of previous antitumor therapy which is CTCAE Grade >1 before the start of study treatment, except for alopecia or hemoglobin greater than or equal to 9.0 g/dL or greater than or equal to 5.6 mmol/L.

Subjects with any clinical condition that is considered unstable or might jeopardize the safety of the subject and/or influence the subjects compliance in the study.

Subjects who have received systemic anticancer therapy within 3 weeks before the start of study treatment. Mitomycin C or nitrosoureas must be excluded within 6 weeks before the start of study treatment.

Subjects who have received radiotherapy to tumor lesions that would be chosen as target lesions (measurable disease) within 4 weeks before the start of treatment, except if there is objective evidence of progression of the lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 between the

prior radiotherapy and the screening computed tomography (CT) or magnetic resonance imaging (MRI) scan. Palliative radiotherapy to nontarget lesions is allowed at the investigators discretion.

Use of drugs that inhibit renal tubular secretion (e.g. probenecid and cimetidine) within 2 weeks before the start of study treatment.

Use of strong cytochrome P450 3A4 (CYP3A4) inhibitors or strong CYP3A4 inducers within 2 weeks before the start of study treatment.

Subjects who have previously received anetumab ravtansine.

Subjects who are concurrently receiving any other investigational agents.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol: Phase 2 Cohort was not performed because we did not accrue at least 6 subjects in the Safety run-in cohort. The first 6 evaluable subjects enrolled in whom the higher of 2 de-escalating doses of anetumab ravtansine will be evaluated in order to determine the recommended Phase 2 dose.
Period: Overall Study
Arm/Group | 1/Safety Run-in Arm
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The highest dose tested at which no more than 1 dose limiting toxicity occurs. A dose limiting toxicity is defined as any treatment emergent adverse event (TEAE) (i.e., absolute neutrophil count <500/mm^3 for ≥7 days) occurring during Cycle 1 and regarded to be at least possibly related to anetumab ravtansine.
Time Frame: 21 days after initiation of study therapy
Population: This outcome measure was not done because the study was terminated due to slow, insufficient accrual.
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Proportion of Subjects Who Experienced a Partial or Complete Response
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). A complete response is disappearance of all target lesions. A partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 6 weeks
Measure: Number; unit: proportion of participants
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 2
proportion of participants
  Partial Response | 0
  Complete Response | 0

3. Secondary Outcome: Progression Free Survival
Description: Length of time from start of treatment to time of progression or death, whichever occurs first. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: At Disease Progression, approximately 6 weeks.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 2
Weeks | 5.5 [5.3 to 5.7]

4. Secondary Outcome: Duration of Response
Description: Duration of Response is from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR). Length of time criteria are met for partial response or complete response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). A complete response is disappearance of all target lesions. A partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: At Disease Progression, approximately 6 weeks from start of treatment
Population: No participant met the criteria for a complete response or partial response.
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Length of time from start of treatment to death from any cause.
Time Frame: At Death, an average of 7.5 weeks after start of first cycle for both patients.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 2
Weeks | 7.6 [5.7 to 9.6]

6. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Participants on the Safety run-in phase was assessed for approximately two months and 5 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Safety Run-in Arm
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Participants on the Safety run-in phase was assessed for approximately two months and 5 days.
Arm/Group | 1/Safety Run-in Arm
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Safety Run-in Arm (N=2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1/Safety Run-in Arm (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3)
Fatigue (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1/1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1/1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02839681/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT02839681/ICF_001.pdf